CLINICAL TRIAL: NCT05318677
Title: The Relationship Between Sensory and Motor Proficiency For Children With Spina Bifida
Brief Title: Sensory and Motor Proficiency For Children With Spina Bifida
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ozden Baskan, Principal Investigator, Pamukkale University
Other Study IDs: OBaskan; AKitis (Other: PamukkaleU)
Record Dates: First submitted 2022-03-24; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Spina Bifida; Sensory Disorder; Motor Disorders; Upper Extremity Dysfunction
Keywords: spina bifida; upper extremity function; sense; motor function
MeSH Terms: conditions — Spinal Dysraphism; Sensation Disorders; Motor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 1: Fifteen patients with spina bifida aged 8-12 years living in Denizli province were included in the study. The participants were informed about the research and read the voluntary consent form, and written consent was obtained from their families since the participants were children.
  Children with literate, well cooperated, aged 8-12 years, and attending any primary school were included in the study. Children who had a second illness and could not be contacted were not included in the study. Non-dominant and dominant extremities of all cases were evaluated by the tests. It was recorded socio-demographic data were questioned. Sensory evaluation forms for upper extremities, Bruininks-Oseretsky motor proficiency, and ability tests were administered by a physiotherapist.
- 2: 20 healthy subjects as a control group aged 8-12 years living in Denizli province were included in the study. The participants were informed about the research and read the voluntary consent form, and written consent was obtained from their families since the participants were children.
  Children with literate, well cooperated, aged 8-12 years, and attending any primary school were included in the study. Children who had a second illness and could not be contacted were not included in the study. Non-dominant and dominant extremities of all cases were evaluated by the tests. It was recorded socio-demographic data were questioned. Sensory evaluation forms for upper extremities, Bruininks-Oseretsky motor proficiency, and ability tests were administered by a physiotherapist.

SUMMARY:
Spina bifida is one of the neural tube defects that cause neuromuscular dysfunction. Spina bifida is a disease accompanied by motor paralysis, musculoskeletal problems, Arnold-Chiari malformation, osteoporosis, hydrocephalus, upper limb coordination disorder. The affected upper extremity functionality and hand skills are very important for independence in daily living activities.

There are some studies in the literature showing that upper extremity motor function is affected in patients with spina bifida. However, no study was found in which the upper extremity was investigated in terms of sensory and motor proficiency.The social and professional aspects of the upper extremity are of great importance.Therefore, our study aims to investigate the effects of upper extremity sensory and motor proficiency in patients with spina bifida

DETAILED DESCRIPTION:
This study aims to examine the relationship between hand skills and upper extremity functional level patients with spina bifida. Fifteen patients with spina bifida and 20 healthy subjects as a control group aged 8-12 years living in Denizli province were included in the study. The participants were informed about the research and read the voluntary consent form, and written consent was obtained from their families since the participants were children.

Children with literate, well cooperated, aged 8-12 years, and attending any primary school were included in the study. Children who had a second illness and could not be contacted were not included in the study. Non-dominant and dominant extremities of all cases were evaluated by the tests. It was recorded socio-demographic data were questioned. Sensory evaluation forms for upper extremities, Bruininks-Oseretsky motor proficiency, and ability tests were administered by a physiotherapist.

All sensory evaluations; In a quiet, bright, warm room with only the physiotherapist and the subject, the evaluation was made while the subject was sitting in a chair with back support.

* Stereognosis: For the evaluation of stereognosis, the subject was asked to recognize the materials placed in his hand by using a pen, paper, clip, cotton, and coin while his visual field was closed. Both dominant and nondominant extremities were evaluated.
* Graphesthesia: When the visual field is closed, square, triangle, circle, and cross signs drawn on the palms of the subjects were asked to know these shapes.
* Finger identification: The patient's fingers were numbered and the patient was asked to know which finger was touched by touching his finger while his visual field was closed, verbally or by showing.
* Kinesthetic sense of hands: A total of 9 evaluations were made, the first of which was a trial, while the patient's visual field was closed. The evaluation was made for both dominant and nondominant extremities. The evaluation was made with both eyes open and closed.8 Evaluation under the title of visual and kinesthetic kinesthesia was scored between 0-3.
* The motor proficiency and ability level of the cases were evaluated with the Bruininks-Oseretsky Test, which is used to evaluate the motor abilities of children aged 4.5-14.5 years in pediatric rehabilitation. The test consists of a total of 46 tests, 8 of which are subtests. Subtests to be applied to the patients in the study: Drawing lines through the path and folding paper tests were performed for the fine motor precision test.

Copying a square and copying star tests were applied for fine motor integration.

Transferring coins has been applied for manual dexterity. The case took the coin with the dominant hand and puts it in the box with the non-dominant hand. The number of coins left in the well in 15 seconds is calculated. The case was given 2 attempts.For upper extremity coordination, the tests of dropping and catching the ball with both hands and dribbling the ball with alternating hands were applied. For the test of dropping and catching the ball with both hands, the subject was given a tennis ball and asked to catch the ball by throwing it on the ground with both hands. A trial was allowed before starting the test.

ELIGIBILITY:
Inclusion Criteria:Children with literate, well cooperated, aged 8-12 years, and attending any primary school were included in the study.

Exclusion Criteria:

* Children who had a second illness and could not be contacted were not included in the study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifteen patients with spina bifida and 20 healthy subjects as a control group aged 8-12 years living in Denizli province were included in the study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sensory assesment of the children | May 2010
  Sensory evaluation in the cases was made by evaluating the senses of stereognosis, graphesthesia, finger identification, and kinesthesia.
Motor proficiency of the children | May 2010
  Motor proficiency of the children was assessed by Bruiniks Oseretsky test.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Baskan, Principal Investigator — Pamukkale University

IPD SHARING:
Plan to Share IPD: No